CLINICAL TRIAL: NCT01080352
Title: Evaluation of Cytotoxicity and Genetic Changes of High Dose Vitamin C Infusions in Castration Resistant Metastatic Human Prostate Cancer
Brief Title: Vitamin C as an Anti-cancer Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-008692-33
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer; palliative care; antioxidants; ascorbic acid; rna expression
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin C treatment (Experimental): Each subjects receive 12 weeks of 1 weekly treatment with intravenous vitamin c.
  5grams are given at week 1, 30 grams at week 2 and 60 grams at week 3-12. If eligibility criteria are met the subject may continue with 1 weekly vitamin c treatment of 60 grams at week 13-20.
  Interventions: Drug: Ascorbic Acid (Vitamin C)

INTERVENTIONS:
Drug: Ascorbic Acid (Vitamin C) — 60grams of ascorbate given intravenous infusion in 1000ml sterile water.

SUMMARY:
Can high dose, intravenous Vitamin C prolong life for patients with metastatic prostate cancer?

Prostate cancer is the most common cancer (excluding skin cancer) in men in Denmark and the Unites States. When metastatic disease is present cure is no longer possible. The main treatment at this stage is castration, either surgical or medical, ending the patients testosterone production and causing a temporary regression in disease activity.

Eventually, the cancer will progress, usually within 2 years from the castration, with a more aggressive course and a survival of 2-3 years.

The current treatment option for the patients, who have undergone castration and have disease progression, is chemotherapy with only limited gains in quality of life and survival.

This clinical study is a phase 2 study to evaluate the effects of high dose intravenous vitamin c in subjects with early castration resistant prostate cancer.

Primary endpoint:

* Prostate specific antigen (PSA) changes after 12 to 20 weekly vitamin c infusions

Secondary endpoints:

* Bone metastases changes after 12 to 20 weekly vitamin c infusions
* Changes in bone specific alkaline phosphates, oxidative DNA-damage, PINP, NTX after 12 to 20 weekly vitamin c infusions
* RNA-expression changes in prostatic tumor tissue after 12 to 20 weekly vitamin c infusions
* RNA-expression changes in lymphocytes after 12 to 20 weekly vitamin c infusions

Tertiary endpoints:

* Pharmacokinetics of vitamin c in the elderly cancer patients

Methods and material:

* 80 subjects are included (efficacy evaluation when 20 subjects have been evaluated for extension arm)
* Each subject receives a weekly infusion of 60 grams vitamin c (in the form of ascorbate) for 12 to 20 weeks

DETAILED DESCRIPTION:
Vitamin C for palliative treatment:

Intravenous vitamin C has been used since the 1970's for terminally ill cancer patients claiming big increases in survival time. The efficacy of the drug is questioned and no randomized, controlled trial of Vitamin C's efficacy on cancer patients survival has been made.

Recent results from in vitro and xenograft studies in mice has shown some promise for vitamin c as a cytotoxic agent against cancer cells.

The following parameters are recorded for baseline:

* Biomarkers (PSA, bALP, NTX, PINP)
* Routine blood work (hgb, creatinine, p-vitamin c etc.)
* Radio nucleotide bone scintigraphy
* Prostate biopsies for later microarray (Affymetrix ST1.0)
* Urine samples 8-oxo-guanine(for oxidative DNA-damage measurements)

These parameters are repeated after treatment, usually after 12 to 26 weeks after the first vitamin c infusion.

ELIGIBILITY:
Inclusion Criteria:

* Castration resistant metastatic prostate cancer (bony or visceral metastases)
* Gleason sum > 6
* PSA > 10 ng/ml
* ECOG < 3
* Prior orchidectomy or LHRH antagonist/agonist treatment
* Must give informed content

Exclusion Criteria:

* Synchronous active cancer (skin cancer excluded)
* Prior chemotherapy
* History of oxalate renal stones
* Glucose-6-phosphate dehydrogenase deficiency
* Impaired renal function (creatinine > 200micromoles/L
* Haemochromatosis
* Cardiac disease (NYHA > 2, CSS > 2, recent AMI (less than 6 months)
* Recent major surgery (less than 4 weeks before inclusion and more than 2 days of admittance time)
* Prior intended curative treatment of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
PSA changes after 12-20 weeks of treatment | 12, 20 and 26 weeks

SECONDARY OUTCOMES:
Bone metastases changes | 12, 26 and 52 weeks
bALP changes | 12, 20, 26 and 52 weeks
NTX changes | 12, 20, 26 and 52 weeks
PINP changes | 12, 20, 26 and 52 weeks
8-oxo-guanine changes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kari J Mikines, MD, DsMC, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Departmen of Urology, Copenhagen University Hospital at Herlev, Herlev, DK, Denmark

REFERENCES:
- [Derived] Nielsen TK, Hojgaard M, Andersen JT, Jorgensen NR, Zerahn B, Kristensen B, Henriksen T, Lykkesfeldt J, Mikines KJ, Poulsen HE. Weekly ascorbic acid infusion in castration-resistant prostate cancer patients: a single-arm phase II trial. Transl Androl Urol. 2017 Jun;6(3):517-528. doi: 10.21037/tau.2017.04.42. PMID 28725594
- [Derived] Nielsen TK, Hojgaard M, Andersen JT, Poulsen HE, Lykkesfeldt J, Mikines KJ. Elimination of ascorbic acid after high-dose infusion in prostate cancer patients: a pharmacokinetic evaluation. Basic Clin Pharmacol Toxicol. 2015 Apr;116(4):343-8. doi: 10.1111/bcpt.12323. Epub 2014 Oct 7. PMID 25220574
- See also: Participant information (in Danish) — http://www.herlevhospital.dk/menu/Afdelinger/Urologisk_Afdeling_H/Forskning/Vitamin+C/